CLINICAL TRIAL: NCT06514105
Title: Effect of High-intensity Laser Therapy on Supraspinatus Tendon Elasticity in Subacromial Impingement Syndrome: A Double-blind Randomized Controlled Study
Brief Title: Effect of High-intensity Laser Therapy on Supraspinatus Tendon Elasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, Esin Akbas, Assistant Professor Dr, Adiyaman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADU-FTR-EA-01
Record Dates: First submitted 2024-07-11; First posted 2024-07-23 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2024-07

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Elasticity Imaging Techniques; Physical Therapy Modalities; Rotator Cuff
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: The study was planned as double-blind, randomized controlled. There are two groups in the study. The groups consist of the control group and high intensity laser group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization will be done by the physiotherapist who applies the physiotherapy program and high-intensity laser. The patient, the measuring radiologist, and the investigator will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High intensity laser group (Active Comparator): In addition to the physiotherapy program, high intensity laser application will be applied to the high intensity laser group.
  Interventions: Other: Physiotherapy program; Other: High intensity laser
- Control group (Active Comparator): In addition to the physiotherapy program, sham high intensity laser application will be applied to the control group.
  Interventions: Other: Physiotherapy program; Other: Sham high intensity laser

INTERVENTIONS:
Other: Physiotherapy program — All patients participating in the study will be included in the physiotherapy program. Physiotherapy program consist of hot-pack (for 15 minutes), ultrasound (Continuous ultrasound, for 5 minutes, 1-MHZ 1.5W/cm2, a 5-cm ultrasound head on the subacromial region),TENS (for 20 minutes with the BTL 4000 combined device) and exercise program (Stretching exercises for the rotator cuff, rhomboid muscles, levator scapula, serratus anterior and pectoaral muscles and strengthening the muscles around the shoulder with a resistance exercise band selected in a color appropriate to the patient's strength).
Other: High intensity laser — High intensity laser will be applied using the BTL-6000 (BTL Company, UK) device. The first 5 sessions will be applied to the painful area by making circular movements from the center to the outside for 100 seconds at a power of 10W and a dose of 10 J/cm2 (analgesic effect). The last 5 sessions will be applied to the painful area with linear movements at 4W power and 100 J/cm2 dose (biostimulation effect) for 10 minutes and 25 seconds.
  Arms: High intensity laser group
Other: Sham high intensity laser — In sham application, the patient will be positioned on the treatment stretcher and the device will be turned on. The guide light of the high-intensity laser device, which gives the same color as the laser light, will be applied to the subacromial region in circular movements from outside to inside and from inside to outside.
  Arms: Control group

SUMMARY:
Subacromial impingement syndrome, one of the most common causes of shoulder pain. In studies investigating the effectiveness of high-intensity laser in patients with subacromial impingement syndrome, it was stated that high-intensity laser reduced the complaints of patients in the early and late periods. However, there is no research examining the effect of high-intensity laser on the supraspinatus tendon. Therefore, the investigators aimed to investigate the effect of high-intensity laser on the supraspinatus tendon using shear wave elastography.

DETAILED DESCRIPTION:
Subacromial impingement syndrome, one of the most common causes of shoulder pain, occurs when the supraspinatus tendon, subacromial bursa or bicipital tendon becomes compressed between the acromion, coracoacromial ligament, coracoid process and/or acromioclavicular joint during shoulder movements. Several factors contribute to subacromial impingement syndrome, including weakening of the rotator cuff, capsular tension, poor scapulohumeral rhythm, and muscular imbalance in the upward rotation force of the scapula. Steroid and non-steroidal anti-inflammatory agents, physiotherapy applications, laser therapy, manual therapy, ESWT and active and passive normal joint movements involving the shoulder joint are frequently applied treatments in the treatment of subacromial impingement syndrome.

It is stated that high-intensity laser treatment can quickly produce photochemical and photothermic effects in deep tissue. Therefore, collagen production in tendons is promoted and blood flow, vascular permeability and cell metabolism can be increased. As a result of all these processes, tissue healing begins and painful stimuli decrease. In studies investigating the effectiveness of high-intensity laser in patients with subacromial impingement syndrome, it was stated that high-intensity laser reduced the complaints of patients in the early and late periods. However, there is no research examining the effect of high-intensity laser on the supraspinatus tendon. Therefore, in this study, the investigators aimed to investigate the effect of high-intensity laser on the supraspinatus tendon using shear wave elastography.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain lasting more than 6 weeks.
* Diagnosed with subacromial impingement
* Being between the ages of 30-60
* Volunteering to participate in the study

Exclusion Criteria:

* Acute inflammatory disease affecting the shoulder area
* Presence of cervical radiculopathy
* Surgical intervention involving the shoulder and neck area
* Soft tissue or bone problems affecting the shoulder
* had any neurologic problems
* Patients who wish to withdraw from the study at any stage after volunteering

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Elasticity Measurement | 2 weeks
  In patients diagnosed with subacromial impingement syndrome as a result of physical examination, the degree of elasticity of the supraspinatus tendon and supraspinatus muscle on the relevant side will be evaluated numerically by Shear Wave elastography. All patients will be scanned by an expert radiologist using a high-resolution broadband linear probe with a Samsung RS 85 Prestige device. While the patients are sitting comfortably and the arm is in a neutral position, the linear probe will be placed parallel to the supraspinatus tendon and the tendon will be displayed in the longitudinal direction. Velocity and elasticity values of the muscle in kPa will be measured using 3 mm diameter range of interest (ROIs) with the help of Shear Wave elastography in the supraspinatus tendon at a distance of 0.5-1.5 cm from the tuberculum majus. For each patient, the measurement will be repeated three times and the average of these three values will be recorded.

SECONDARY OUTCOMES:
Functional level | 2 weeks
  The functional level of the shoulder will be evaluated with the Shoulder Pain and Disability Scale. This scale consists of a total of 13 questions, where each question is scored between 0-10. The scores from the first 5 questions measure the pain level out of 50, and the scores from the next 8 questions measure the disability level out of 80. A high score from the scale indicates a high level of pain and disability.
Pain assessment | 2 weeks
  The severity of patients' shoulder pain will be evaluated with a visual analog scale (VAS). VAS: The left end of a 10 cm straight line represents no pain, and the right end represents unbearable pain. The patient will be asked to mark the pain he feels on the VAS scale during the test, and then this value will be measured and recorded with the help of a ruler.

CONTACTS AND LOCATIONS:
Overall Officials: Esin Akbaş, Principal Investigator — Adiyaman University
Locations (1):
- Adiyaman university, Adıyaman, Adıyaman Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No